CLINICAL TRIAL: NCT05295056
Title: Clinical Performance of the AFGen1 Device Over a 7-day Period
Status: Completed | Type: Observational
Sponsor: TriVirum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AFib-Chek-001
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Afib; Irregular Heart Beat; Arrhythmias, Cardiac; Arrhythmia Atrial; Arrhythmias Paroxysmal; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Permanent atrial fibrillation: Known to have permanent atrial fibrillation
  Interventions: Device: AFGen1 Device Wear Test
- Healthy control: Healthy controls
  Interventions: Device: AFGen1 Device Wear Test; Device: AFGen 1 Device Single Use

INTERVENTIONS:
Device: AFGen1 Device Wear Test — Participant wears the device for 7 days
Device: AFGen 1 Device Single Use — Participant wears the device in conjunction with a standard ECG
  Groups: Healthy control

SUMMARY:
AFGen1 is indicated for use on symptomatic or asymptomatic adults who are at risk of developing or who have atrial fibrillation, where a software assisted analysis of ambulatory ECG is needed to identify episodes of Afib. The purpose of this study is to establish the clinical performance of the AFib-Chek device (a.k.a. Device) on human participants.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate that the ECD signal acquired by the AFGen1 device is as of adequate quality and is suitable to support its intended use for the detection of AFib.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ willing to sign the consent form

Exclusion Criteria:

1. Implanted pacemakers
2. Implanted cardioverter defibrillators
3. Implanted cardiac resynchronization devices
4. Potential life-threatening arrythmias
5. Physical or mental health conditions that would prevent the person from being able to follow instruc-tions regarding participation in the study
6. Open wounds, abraded or irritated skin at the application site
7. Planned to undergo a MRI during the course of the study duration

Ages: 65 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: The study shall involve approximately 30-50 participants (approximately equal number of males and females, equal number with BMI < and > 35) meeting inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Quantitative Evaluation | 7 days
  For the quantitative evaluation of the mean and standard deviation of the QRS correlations for all study subjects and for the end of the wear period for those relevant subjects, the mean cor- relation coefficient must be greater than 0.95 and standard deviation must be less than 0.05 to validate a 95% confidence interval with significant factor of assurance.
Qualitative Equivalence Evaluation | 7 days
  For the qualitative equivalence evaluation according to the two cardiologists the confirmation of equivalence must be greater than 95%.
Adhesive performance | 7 days
  For the adhe sive performance element of the stud y; t he overall average wear time for the de- vice must be greater than 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No